CLINICAL TRIAL: NCT01006811
Title: Efficacy and Tolerability of the Modified Atkins Diet in Patients With Infantile Spasms: a Pilot Study.
Brief Title: Use of the Modified Atkins Diet in Infantile Spasms
Acronym: ADIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr Suvasini Sharma, All India Institute of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADIS
Record Dates: First submitted 2009-11-01; First posted 2009-11-03 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Infantile Spasms
Keywords: West syndrome; Hypsarrhythmia
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- modified Atkins diet (Experimental)
  Interventions: Dietary Supplement: modified Atkins diet; Other: modified Atkins diet

INTERVENTIONS:
Dietary Supplement: modified Atkins diet — Modified Atkins Diet administration
  1. Carbohydrates intake restricted to 10 grams/ day. (Carbohydrate values of various food items will be explained in detail, and exchange lists provided. Four 2.5 grams carbohydrate exchange items will be allowed in a day.)
  2. Fats (e.g. cream, butter, oils, ghee) encouraged.
  3. Proteins (cheese, fish, eggs, chicken, soya products) unrestricted.
  4. Clear carbohydrate-fluids not restricted.
  5. Calcium and multivitamin supplementation will be provided.
  Other Names: Dietary treatment
Other: modified Atkins diet — Modified Atkins Diet administration
  1. Carbohydrates intake restricted to 10 grams/ day. (Carbohydrate values of various food items will be explained in detail, and exchange lists provided. Four 2.5 grams carbohydrate exchange items will be allowed in a day.)
  2. Fats (e.g. cream, butter, oils, ghee) encouraged.
  3. Proteins (cheese, fish, eggs, chicken, soya products) unrestricted.
  4. Clear carbohydrate-fluids not restricted.
  5. Calcium and multivitamin supplementation will be provided.
  Other Names: Dietary treatment

SUMMARY:
Infantile spasms constitute a type of catastrophic epilepsy syndrome occuring in young children. The ketogenic diet has been shown to be very effective in these children. The modified Atkins diet is a less restrictive option than the ketogenic diet, which has been effective in preliminary studies on refractory epilepsy in children, adolescents and adults. Modified Atkins diet may be of special importance in infants, as proteins are not restricted, hence no problems with growth are expected. Hence this pilot study has been planned to evaluate the efficacy and tolerability of the modified Atkins diet in infantile spasms refractory to conventional treatment (ACTH, vigabatrin, and anti-epileptic drugs).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6 months to 3 years.
2. Presence of epileptic spasms in clusters, with electroencephalographic evidence of hypsarrhythmia or its variants), having at least one cluster per day.
3. Treatment with at least corticosteroid/ ACTH or Vigabatrin and one other AED( sodium valproate, pyridoxine, topiramate, zonisamide, benzodiazepines (clobazam, clonazepam, nitrazepam).

Exclusion Criteria:

1. Known or suspected inborn error of metabolism, as evidenced by: Clinical suspicion of metabolic disorder as evidenced by 2 or more of the following- a history of parental consanguinity, prior affected siblings, unexplained vomiting, intermittent worsening of symptoms, recurrent episodes of lethargy, altered sensorium, or ataxia, hepatosplenomegaly on examination And/ or 2 or more of the following biochemical abnormalities High blood ammonia (>80mmol/L), High arterial lactate (>2 mmol/L), metabolic acidosis (pH <7.2), hypoglycaemia (blood sugar <40 mg/dl), abnormal urinary aminoacidogram, presence of reducing sugars or ketones in urine, and positive results on urine neurometabolic screening tests.
2. Motivational or psychosocial issues in the family which would preclude compliance
3. Systemic illness- chronic hepatic, cardiac, renal or pulmonary disease

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
seizure reduction as per parental reports | 3 months
  seizure control at the end of 3 months will be classified as: spasm free; > 50% reduction in spasms; and < 50% reduction in spasms

SECONDARY OUTCOMES:
adverse effects of the diet as per parental reports | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Suvasini Sharma, MD, DM, Principal Investigator — All India Institute of Medical Sciences; Sheffali Gulati, MD, Study Director — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Sharma S, Sankhyan N, Gulati S, Agarwala A. Use of the modified Atkins diet in infantile spasms refractory to first-line treatment. Seizure. 2012 Jan;21(1):45-8. doi: 10.1016/j.seizure.2011.08.009. Epub 2011 Sep 14. PMID 21920781